CLINICAL TRIAL: NCT05665985
Title: Effect Of Moringa Leaf Extract On Disease Activity In Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, Head of Hospital Research Unit, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAP01
Record Dates: First submitted 2022-11-26; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — flocculant protein MO 2.1, Moringa oleifera

STUDY DESIGN:
Intervention Model Description: This study was a Randomized Controlled Trial (RCT) with 30 research samples divided into two groups, containing 15 samples each for the treatment group and 15 for the control group. The treatment group was given Moringa oleifera extract of 40.50 mg/KGBW/day, while the control group was given a placebo for 30 days. The degree of disease activity (DAS28-CRP, DAS28-LED) was assessed before and after the intervention. Intervention with Dry Extract of Moringa Oleifera (trade name is Keloreena Ⓡ , registered number in National Food and Drug Registry: 193332021) The dose given is 1000 mg bi in day for 30 days. Inclusion criteria are Female patients, 18-60 years, who met the RA criteria according to the ACR / EULAR 2010 and VAS> 3. Exclusion criteria are Pregnant, using Methylprednisolone> 8 mg per day, using NSAIDs, and having comorbidities
Who Masked: Participant, Investigator
Masking Description: The capsule form between the drug and the placebo was the same, there was no drug name label on the drug packaging, and only a number was given on the drug packaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa Oliefera (Experimental): Intervention with Dry Extract of Moringa Oleifera (trade name is Keloreena Ⓡ , registered number in National Food and Drug Registry: 193332021) The dose given is 1000 mg bi in day for 30 days.
  Interventions: Drug: Moringa Oleifera
- Placebo (Placebo Comparator): Capsules similar to moringa oliefera, which contain powder, have no pharmacological effect.
  Interventions: Drug: Moringa Oleifera

INTERVENTIONS:
Drug: Moringa Oleifera — Intervention with Dry Extract of Moringa Oleifera (trade name is Keloreena Ⓡ , registered number in National Food and Drug Registry: 193332021) The dose given is 1000 mg bi in day for 30 days.

SUMMARY:
Intervention therapy study of moringa oliefera extract on the degree of activity of rheumatoid arthritis patients. The research subjects were patients with rheumatoid arthritis-intervention with moringa oliefera for 30 days.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a progressive autoimmune disease. Delay in therapy and delay in remission will result in disability. This study is a randomized clinical trial using a new drug for rheumatoid arthritis, moringa oliefera. The choice of moringa oliefera was due to the ability of moringa oliefera in anti-inflammatory and immunosuppressant terms. This drug has also been proven in experimental studies on rheumatoid arthritis animals. This study with 30 research samples divided into two groups, containing 15 samples each for the treatment group and 15 for the control group. The treatment group was given Moringa oleifera extract of 40.50 mg/KGBW/day, while the control group was given a placebo for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA criteria according to the ACR / EULAR 2010
* Visual analog score of more than three.

Exclusion Criteria:

* Pregnancy
* Using Methylprednisolone> 8 mg per day
* Using NSAIDs
* Chronic Kidney Disease
* Diabetes Mellitus
* Heart Failure
* Lever disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
DAS-28 CRP | pre and post intervention (30 day)
  The change of Disease activity score in Rheumatoid arthritis patients
DAS-28 ESR | pre and post intervention (30 day)
  The change of Disease activity score in Rheumatoid arthritis patients

CONTACTS AND LOCATIONS:
Locations (1):
- RS UNS (Universitas Sebelas Maret Hospital), Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No